CLINICAL TRIAL: NCT03527966
Title: rhBMP-2 Versus Vivigen, a Novel Cellular Allograft, in Lumbar Fusion Procedures: a Prospective Randomized Controlled Study
Brief Title: rhBMP-2 Versus Vivigen in Lumbar Fusion Procedures
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: PI left the institution
Sponsor: Virtua Health, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB G17008
Record Dates: First submitted 2018-05-04; First posted 2018-05-17 (Actual); Results first posted 2019-08-07 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Lumbar Spine Degeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: The surgical team, including the surgeons, will be blinded to the treatment options until decompression/instrumentation have been completed. The patients and all staff, including hospital nursing staff, case management, and physical therapists, will be blinded as to which bone graft treatment the patient received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention group - 5cc Vivigen and local autograft (Active Comparator)
  Interventions: Biological: 5cc Vivigen and local autograft
- Control group - small kit rhBMP-2 with local autograft (Active Comparator)
  Interventions: Biological: Small kit rhBMP-2 with local autograft

INTERVENTIONS:
Biological: 5cc Vivigen and local autograft — The single level lumbar instrumented fusion patients assigned to this group will receive 5cc Vivigen and local autograft
  Arms: Intervention group - 5cc Vivigen and local autograft
Biological: Small kit rhBMP-2 with local autograft — The single level lumbar instrumented fusion patients assigned to this group will receive small kit rhBMP-2 with local autograft
  Arms: Control group - small kit rhBMP-2 with local autograft

SUMMARY:
This study is aimed at comparing the overall efficacy (clinical and radiographic) of Vivigen, a novel cellular allograft product, and rhBMP-2 when utilized in lumbar fusion procedures.

DETAILED DESCRIPTION:
The purpose of this study is to compare the overall efficacy (clinical outcome and radiographic fusion) of Vivigen (cellular allograft product) and rhBMP-2 in patients who undergo a single level lumbar instrumented fusion. Specifically, when compared to their control group counterparts treated to rhBMP-2, we hypothesize that the intervention group administered Vivigen would, following surgery, experience:

1. Comparable mean postoperative leg/back pain score, where the pain scores are obtained using the numeric rating scale of 0-no pain, to 10-worst pain possible
2. Comparable inpatient length of stay (LOS)
3. Comparable postoperative Oswestry Disability Index (ODI) score (0-no disability, to 100-maximum disability possible), two weeks, 6 weeks, 3 months, 6 months, and 1 year postoperatively
4. Comparable fusion rates, evaluated via CT scan I year postoperatively

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older;
2. Diagnosed with lumbar degenerative/isthmic spondylolisthesis, degenerative disc disease with axial low back pain and neurologic symptoms, failed conservative treatment and eligible for a single level lumbar instrumented fusion;
3. Willing to provide informed consent, participate in study, and comply with study protocol.

Exclusion Criteria:

1. Pregnant or contemplating pregnancy prior to surgery;
2. Serious spinal conditions (e.g. spinal cord compression, cauda equina syndrome, spinal infection, spinal tumor, spinal fracture, inflammatory or systemic spinal arthritis);
3. Surgery involving more than 2 vertebral levels;
4. Worker's compensation or personal injury related to lumbar spine (treatment outcomes may be affected by patient's personal interests; could also run into potential issues with reimbursement).
5. Lactating women
6. Patients who have a known or suspected allergy to Gentamicin Sulfate, Meropenem, Vancomycin, Dimethyl Sulfoxide (DMSO), and Human Serum Albumin
7. Immune compromised patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2018-07-27 (Actual); Study Completion 2018-07-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Virtua Memorial Hospital, Mount Holly, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Plan to disseminate study findings via conference representation and journal publication using de-identified analyzed data

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Group - 5cc Vivigen and Local Autograft | Control Group - Small Kit rhBMP-2 With Local Autograft
Started | 3 | 0
Completed | 0 | 0
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 3 | 0

BASELINE CHARACTERISTICS:
Population: Study was terminated early when PI left the practice. Three patients were randomized to the intervention group. Zero were randomized to the control group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group - 5cc Vivigen and Local Autograft | Control Group - Small Kit rhBMP-2 With Local Autograft | Total
Number analyzed (Participants) | 3 | 0 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 2
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Full Range); unit: years] | 53 [46 to 65] |  | 52.6 [46 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 |  | 1
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 2 |  | 2
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Oswestry Disability Index (ODI) Score
Description: The ODI is one of the most commonly utilized condition-specific measures of disability used in the management of spinal disorders (0-no disability, to 100-maximum disability possible)
Time Frame: Up to 1 year post surgery
Population: Patients did not attend every follow up visit and then were ultimately lost to follow up. Study was also terminated early when the PI left his practice so on patients were never randomized in the control group.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Intervention Group - 5cc Vivigen and Local Autograft | Control Group - Small Kit rhBMP-2 With Local Autograft
Number analyzed (Participants) | 3 | 0
score on a scale
  ODI at Two weeks: number analyzed (Participants) | 2 | 0
  ODI at Two weeks | 78.5 [70 to 87] |
  ODI at Six weeks: number analyzed (Participants) | 2 | 0
  ODI at Six weeks | 42 [26 to 58] |
  ODI at Three months | 36.6 [8 to 70] |
  ODI at Six months: number analyzed (Participants) | 1 | 0
  ODI at Six months | 36 [36 to 36] |
  ODI at 1 year: number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Mean Postoperative Leg/Back Pain Score
Description: Pain scores are obtained using the numeric rating scale of 0-no pain, to 10-worst pain possible
Time Frame: Average of 3 days in hospital
Population: Study was terminated early before any patients were randomized to the control group.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Intervention Group - 5cc Vivigen and Local Autograft | Control Group - Small Kit rhBMP-2 With Local Autograft
Number analyzed (Participants) | 3 | 0
score on a scale | 5.3 [0 to 10] |

3. Secondary Outcome: Mean Inpatient Length of Stay
Time Frame: Average of 3 days in hospital
Population: The study was terminated early before any patients were randomized to the control group.
Measure: Mean (Full Range); unit: days
Arm/Group | Intervention Group - 5cc Vivigen and Local Autograft | Control Group - Small Kit rhBMP-2 With Local Autograft
Number analyzed (Participants) | 3 | 0
days | 1 [1 to 1] |

4. Secondary Outcome: Fusion Rates, Evaluated Via CT Scan I Year Postoperatively
Time Frame: 1 year post surgery
Population: No patient returned for their 1 year post op scan
Arm/Group | Intervention Group - 5cc Vivigen and Local Autograft | Control Group - Small Kit rhBMP-2 With Local Autograft
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: Zero participants in the control group were at risk for all-cause mortality, serious adverse events, and other (not including serious) adverse events as the study was terminated early before any patients enrolled in that study arm. Adverse events collected per clinicaltrials.gov definitions. Protocol considered opioid related adverse events (ORAEs) an area of special interest but none were reported.
Arm/Group | Intervention Group - 5cc Vivigen and Local Autograft | Control Group - Small Kit rhBMP-2 With Local Autograft
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/0
Other Adverse Events (participants affected / at risk) | 0/3 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-08): https://cdn.clinicaltrials.gov/large-docs/66/NCT03527966/Prot_SAP_000.pdf